CLINICAL TRIAL: NCT00221338
Title: Clinical Trial of Gabapentin to Decrease Postoperative Delirium and Pain in Surgical Patients
Brief Title: Clinical Trial of Gabapentin to Decrease Postoperative Delirium and Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H5636-26795-01
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Delirium; Postoperative Pain; Opioid Use; Hospital Length of Stay
Keywords: gabapentin; pain; surgery; delirium; cognitive decline
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative; Pain; Delirium; Cognitive Dysfunction | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Experimental): Double blind, placebo controlled
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Double blind
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — This is a Double blind, placebo-controlled experimental study in which gabapentin adjusted for renal clearance (or placebo) is given preoperatively and also the first three postoperative days
  Other Names: gabapentin versus placebo

SUMMARY:
This will be a double blind, placebo-controlled study of patients ≥65 years of age undergoing surgery of the spine, hips and knees replacement at the University of California, San Francisco (UCSF) Medical Center. Intraoperative anesthetic and postoperative pain management will be standardized. Patients will be randomized to receive either placebo or gabapentin preoperatively, and continued postoperatively until discharge. Intraoperative anesthetic and other postoperative pain management strategies will be standardized. Postoperative delirium will be measured using structured interviews. Cognitive function will be measured using a battery of neurocognitive tests pre- and post-operatively. Using an intention to treat strategy, we, the researchers at UCSF, will compare the incidence of postoperative delirium and cognitive dysfunction, the amount of postoperative pain, and narcotic requirements between the two groups. The primary outcome will be postoperative delirium. Secondary outcomes will be postoperative pain and opioids use, and length of hospital stay, and cognitive dysfunction.

DETAILED DESCRIPTION:
Postoperative delirium is a common condition, occurring in 10-70% of surgical patients after major surgery. To date, few studies have examined events in the postoperative period as contributing factors to postoperative delirium. We recently completed a study in over 500 geriatric surgical patients to examine whether the mode of postoperative analgesia delivery, medication types, and the severity of postoperative pain may impact the occurrence of postoperative delirium. In this study, 46% of patients developed postoperative delirium on either the first or second postoperative day. By multivariate logistic regression, variables which had independent association with postoperative delirium included age ≥80 years, moderate to severe preoperative resting pain, and increased level of resting pain postoperatively in comparison with preoperative baseline. When the analysis was focused on patients who used Patient Controlled Analgesia (PCA) alone for postoperative pain control, the amount of narcotic used (hydromorphone) was significantly higher in those with postoperative delirium as compared to those without, suggesting that inadequate pain control and/or the central effects of opioids may be associated with postoperative delirium. Since increasing the doses of opioids in the elderly patients will likely lead to unwanted side effects such as respiratory depression, the addition of a non-opioid agent may result in a narcotic-sparing effect, and also reducing pain postoperatively.

Gabapentin is a structural analog of gamma-amino butyric acid, and has been used as an anti-convulsant and anti-nociceptive drug. It is not metabolized in humans (therefore no hepatic enzyme induction), and is eliminated from the body by renal clearance. In animal studies, gabapentin has been demonstrated to be effective in reducing both allodynia and hyperalgesia, and may have selective effect on the nociceptive process involved in central sensitization. Gabapentin has been successfully used in the treatment of neuropathic pain and other painful conditions. Recently, there is substantial evidence to suggest that gabapentin also may be useful in the treatment of postoperative pain. To date, there have been nine randomized clinical trials of gabapentin versus placebo including a total of over 700 patients. Taken together, these studies reported that gabapentin given perioperatively significantly reduced postoperative analgesic requirements, and had minimum side effects. The only reported significant side effects in these trials were mild sedation in two studies. In patients with epilepsy, gabapentin can be introduced at therapeutic doses, and presents no safety or serious side effect issues. Since gabapentin has negligible protein binding, it has no interactions with other medications. It is recommended that metabolic and laboratory monitoring is not necessary, and excellent cognitive profile is evident. At UCSF, gabapentin has been used safely in a relatively large number of patients on an empiric bases in the postoperative period, typically in surgical patients with substantial chronic pain, and more recently, in patients who have undergone spinal surgery as an adjuvant agent to narcotics to relieve postoperative radicular pain (personal communication with Peter Koo, Clinical Pharmacist at UCSF). Typically, patients are started on gabapentin 300 mg po TID on the first day, rapidly escalating to 600 mg TID on the second day, and finally to 900 mg TID the third day until discharge. The UCSF experience suggests that gabapentin is well tolerated with minimal side effects.

Hypothesis

We hypothesize that intensive pain management postoperatively using an adjuvant agent, gabapentin, will lead to a decrease in the amount of postoperative pain experienced, thereby resulting in a decrease in the incidence of postoperative delirium in older patients undergoing noncardiac surgery.

Our specific aims were to: 1. Assess whether the administration of gabapentin was associated with decreased occurrence of delirium, 2. Determine the extent to which gabapentin-associated reductions in pain and/or opiate use reduced the occurrence of delirium, and 3. Determine whether the administration of gabapentin was associated with shorter hospital stays. We hypothesized that intensive pain management postoperatively using an adjuvant agent, gabapentin, would lead to a decrease in the amount of opioids received, a decrease in postoperative pain experienced, thereby resulting in a decrease in the incidence of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥65 years of age undergoing surgery involving the spine, hip or knee replacement.
* English speaking.
* Anticipated to stay in the hospital for at least 48 hours.

Exclusion Criteria:

* Patients who take gabapentin preoperatively, or have known sensitivity to the drug, or those unable to be randomized to receive gabapentin.
* Subjects who are unable to provide informed consent.
* Patients with a history of narcotic tolerance.
* Patients with planned two stage spinal procedures (anterior-posterior spinal fusion to be done on two separate days).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 750 (Actual)
Dates: Start 2006-01; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline M Leung, MD, MPH, Principal Investigator — University of California, San Francisco, CA, USA
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share undecided

REFERENCES:
- [Background] Leung JM, Sands LP, Chen N, Ames C, Berven S, Bozic K, Burch S, Chou D, Covinsky K, Deviren V, Kinjo S, Kramer JH, Ries M, Tay B, Vail T, Weinstein P, Chang S, Meckler G, Newman S, Tsai T, Voss V, Youngblom E; Perioperative Medicine Research Group. Perioperative Gabapentin Does Not Reduce Postoperative Delirium in Older Surgical Patients: A Randomized Clinical Trial. Anesthesiology. 2017 Oct;127(4):633-644. doi: 10.1097/ALN.0000000000001804. PMID 28727581
- [Result] Leung JM, Sands LP, Rico M, Petersen KL, Rowbotham MC, Dahl JB, Ames C, Chou D, Weinstein P. Pilot clinical trial of gabapentin to decrease postoperative delirium in older patients. Neurology. 2006 Oct 10;67(7):1251-3. doi: 10.1212/01.wnl.0000233831.87781.a9. Epub 2006 Aug 16. PMID 16914695

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 374 | 376
Completed | 350 | 347
Not Completed | 24 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 350 | 347 | 697
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 350 | 347 | 697
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (6) | 72 (6) | 73 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193 | 158 | 351
  Male | 157 | 189 | 346
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 323 | 315 | 638
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 27 | 32 | 59
Region of Enrollment [Number; unit: participants]
  United States | 350 | 347 | 697
Preoperative Cognitive Status as measured by Telephone Interview for Cognitive Status [Mean (Standard Deviation); unit: units on a scale] — The Telephone Interview For Cognitive Status (TICS) is a standardized, 41-point measure of cognitive function. TICS has been developed and validated as an alternative to the Mini Mental State Examination (MMSE) but, unlike the latter, can be administered either in-person or by telephone. Higher scores means higher cognitive functioning. Lower scores means lower cognitive functioning.
  units on a scale | 34.5 (3.5) | 34.5 (3.1) | 34.5 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Delirium by Study Group
Description: Number of subjects who developed postoperative delirium, as measured by the Confusion Assessment Method, a validated tool for assessing delirium based on DSM-III-R, on any of the first three postoperative days.
Time Frame: postoperative days 1, 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 350 | 347
Participants | 84 | 72

2. Secondary Outcome: Median Postoperative Opioid Doses Across Study Follow up Period
Description: Postoperative intravenous opioid doses converted to morphine equivalents. Median derived from total opioid doses on first, second and third postoperative days.
Time Frame: Study follow up period: postoperative days 1, 2 and 3
Measure: Median (Inter-Quartile Range); unit: morphine equivalents, mg
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 350 | 347
morphine equivalents, mg | 6.7 [1.3 to 20] | 6.7 [2.7 to 24.8]

3. Secondary Outcome: Hospital Length of Stay
Time Frame: Typically within the first week after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 350 | 347
days | 4.4 (3.4) | 4.1 (2.3)

4. Secondary Outcome: Postoperative Pain Score - Postoperative Day 1
Description: Postoperative pain as measured by Visual Analog Pain scale (0=no pain, 10=worst pain imaginable).
Time Frame: Postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 350 | 347
score on a scale | 4 (3) | 4 (3)

5. Secondary Outcome: Postoperative Pain Score - Postoperative Day 2
Description: Postoperative pain as measured by Visual Analog Pain scale (0=no pain, 10=worst pain imaginable).
Time Frame: Postoperative day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 335 | 343
score on a scale | 3 (3) | 4 (3)

6. Secondary Outcome: Postoperative Pain Score - Postoperative Day 3
Description: Postoperative pain as measured by Visual Analog Pain scale (0=no pain, 10=worst pain imaginable).
Time Frame: Postoperative day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 299 | 291
score on a scale | 3 (3) | 3 (3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the time period of 1 year.
Description: In-hospital course was examined daily until discharge for occurrence of postoperative outcomes. All serious adverse events (both anticipated and unanticipated) were reported to the University of California San Francisco Committee on Human Research, and National Institutes of Health (San Francisco, California).
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/350 | 1/347
Serious Adverse Events (participants affected / at risk) | 31/350 | 44/347
Other Adverse Events (participants affected / at risk) | 42/350 | 67/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=350) | Placebo (N=347)
Atrial Flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 6 (6) | 7 (7)
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Heart Block (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Unspecified Dysrhythmia (Cardiac disorders) | 2 (2) | 4 (4) — Charted as "dysrhythmia" or "arrhythmia"
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 4 (4) | 4 (4)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Tachy/Brady (Cardiac disorders) | 4 (4) | 3 (3) — Sinus tachycardia or bradycardia
Hypoxia/Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Reproductive system and breast disorders) | 1 (1) | 3 (3) — Partial or complete collapse of part of or the entire lung
Reintubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acute Renal Failure (Renal and urinary disorders) | 6 (6) | 7 (7) — Requiring new dialysis or acute increase in blood creatinine levels
Acute Infection (Infections and infestations) | 4 (4) | 7 (7) — As evidenced by positive lab cultures
Cerebrovascular accident (Vascular disorders) | 2 (2) | 0 (0) — Stroke or TIA shown by MRI
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 3 (3)
Reoperation (Surgical and medical procedures) | 2 (2) | 2 (2) — Requiring unscheduled second procedure within same hospital stay
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Esophageal Tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — "Mallory-Weiss tear," nasogastric tube placed for 24 hours and tear resolved, advancing to regular diet.
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Anterior dislocation of left hip, closed reduction on floor without complication. Occurred twice on POD5 and POD7.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=350) | Placebo (N=347)
Oxygen Desaturation (Respiratory, thoracic and mediastinal disorders) | 37 (37) | 56 (56) — Oxygen desaturation below 95% but higher than 88%, as measured by pulse oximetry.
Sedation (Nervous system disorders) | 3 (3) | 6 (6) — Median sedation as defined as RASS score -2 (light sedation) or -3 (moderate sedation)
Syncope (General disorders) | 0 (0) | 5 (5)
Dysphagia (General disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Orthostatic Hypotension (General disorders) | 1 (1) | 1 (1)
Dizziness (General disorders) | 1 (1) | 2 (2)
Nausea (General disorders) | 1 (1) | 1 (1)
Hallucinations (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No